CLINICAL TRIAL: NCT05647525
Title: Sichuan Academy of Medical Sciences - Sichuan Provincial People's Hospital
Brief Title: The Etiology of New-onset Status Epilepticus
Status: Completed | Type: Observational
Sponsor: Jie Liu (Other)
Responsible Party: Sponsor-Investigator, Jie Liu, Professor, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Other Study IDs: Liujiessy
Record Dates: First submitted 2022-12-04; First posted 2022-12-12 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- status epilepticus with autoimmune encephalitis; status epilepticus without autoimmune encephalitis: To study the relationship between autoimmune-related antibody titres and prognosis during the six-month follow-up
  Interventions: Diagnostic Test: Perform autoimmune encephalitis titer tests

INTERVENTIONS:
Diagnostic Test: Perform autoimmune encephalitis titer tests — We only follow up without intervention.
  Other Names: We only follow up without intervention.

SUMMARY:
This study will help to identify the causes of new epilepsy and provide a basis for the development of a rational and standardized diagnosis and treatment plan to reduce the rate of disability and death.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Status Epilepticus
* Sign the informed consent form

Exclusion Criteria:

* Patients with previous epilepsy
* Missing information such as basic information and treatment history
* Long-term smoking, alcohol and drug abuse
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were selected strictly according to the inclusion and exclusion criteria from January 2021 to December 2022 at Sichuan Academy of Medical Sciences. Inpatient NOSE patients at Sichuan Provincial People's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Death | 2021-12--2022-12

CONTACTS AND LOCATIONS:
Locations (1):
- Jie Liu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided